CLINICAL TRIAL: NCT01576796
Title: Phase II Study of the Efficacy and Safety of a Radiotherapy Dose Complement in the Treatment of Hypoxic Lesions Identified by F-miso PET/CT in Patients With Stage III Non-small-cell Lung Cancer (NSCLC) Not Amenable to Curative Surgical Resection Who Are Candidate for Curative Radio-chemotherapy
Brief Title: Radiotherapy Dose Complement in the Treatment of Hypoxic Lesions Patients With Stage III Non-small-cell Lung Cancer
Acronym: RTEP-5
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHB11-01
Record Dates: First submitted 2012-04-11; First posted 2012-04-12 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Stage III Non-small-cell Lung Cancer
Keywords: Radiotherapy; Fmiso; FDG PETSCAN; FMISO PETSCAN; complement dose; lung cancer; NSCLC; hypoxic lesion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radiotherapy — No additional dose (patients negative F-miso)
  * Radiation therapy is conducted under standard conditions of conformal radiotherapy:
  * The total dose was 66-70 Gy delivered in daily fractions of 2 Gy, 5 days a-week
  With additional dose (patients positive for F-miso)
  The dose in the PTVmiso increased until the maximum tolerable radiation by the lung.

SUMMARY:
This study will assess the efficacy and safety of a radiotherapy dose complement (boost) in the treatment of hypoxic lesions, measured by F-miso PET/CT, in patients with stage III NSCLC not amenable to surgery and candidate for chemoradiotherapy.

Preliminary studies in head and neck cancers have demonstrated the feasibility and support the medical benefit of this novel approach.

The aim of the study is to assess the efficacy and safety of a radiotherapy dose complement (boost) in this difficult medical condition for which only limited treatment options are available.

DETAILED DESCRIPTION:
Background This phase II study will assess the efficacy and safety of a radiotherapy dose complement (boost) in the treatment of hypoxic lesions, measured by F-miso PET/CT, in patients with stage III NSCLC not amenable to surgery and candidate for chemoradiotherapy.

There is a strong theoretical rationale supporting a radiotherapy dose increase in patients with hypoxic pulmonary tumour. F-miso PET enables in vivo identification and localisation of hypoxic tumoral areas, which constitute a target for an increased total dose of radiation therapy. Preliminary studies in head and neck cancers have demonstrated the feasibility and support the medical benefit of this novel approach. To date, no studies investigating non-small-cell lung cancer patients have been performed.

Given the methodological constraints, we propose a Gehan plan optimizing the number of subjects to be enrolled and the budget.

The project team has been working on imaging of radiotherapy targets for NSCLC for many years within a research group identified by the French National Cancer Institute (INCa) in 2005, and part of the axis 3 of Northwest Canceropole (Prof. Gregoire - Prof. Lartigau - Prof. Vera)2. This project was presented at an EORTC meeting "Imaging and radiotherapy" (organised by Dr. Nestlé) on May 28th 2010. It has been approved by the President of ESTRO (Prof. Gregoire) and the members of SFMN (French Society of Nuclear Medicine) and of the SFRO (French Society of Radiation Oncology) during an "Imaging and Hypoxia" Meeting in September 8th, 2010.

The aim of the study is to assess the efficacy and safety of a radiotherapy dose complement (boost) in this difficult medical condition for which only limited treatment options are available.

Objective(s) of the clinical study Main objective: to evaluate the rate of local control after dose complement in hypoxic lesions [maximum dose without the fraction of total lung volume receiving more that 20 Gy exceeding 30% of the lung (V20)], as determined by F-miso PET/CT.

Secondary objectives:

* 3 months and 1 year toxicity
* Percentage of patients for whom the RT dose could be increased
* Simultaneous variation of the glucose metabolism and hypoxia during radiotherapy
* Predictive value on 1-year survival probability of the variations in glucose metabolism and hypoxia during radiotherapy

Main inclusion criteria

* Patients with stage III non-small-cell lung cancer candidate for curative radio-chemotherapy
* The final inclusion is granted after completion of a dosimetric study confirming that the dose objectives (minimum dose of 60 Gy in 99% of target volume) and constraints to organs at risk can be achieved.

Main assessment criteria

- Percentage of local control as evaluated by CT (RECIST criteria) and FDG PET/CT at 3 months

Assessment criteria for hypoxia Visual analysis: centralized via SFMN net with 3 blinded readers within 8 days (Richin, JCO 2006). Definition of hypoxia and decision about boost dose.

Quantitative analysis: hypoxic fraction determined retrospectively (secondary endpoints and ancillary study). The Gross Target Volume (GTV) will be delineated on FDG PET/CT images using an adaptive method (Vauclin, PMB 2009). The contour of the GTV will be copied onto F-miso PET images after registration. Voxels with a signal to noise ratio greater than 1.2 will be considered as the hypoxic volume.

Experimental plan Assumption: to increase the local control rate at 3 months from 17% to 40%. A two-staged Gehan plan will be implemented. The assumption of therapeutic efficacy is π = 0.4 - In the first stage, 6 patients will receive a radiotherapy dose boost on the hypoxic lesions. If no local control is observed in these 6 patients, the trial will be stopped (power 0.95). In a second stage, the number of patients to be included will be determined according to the number of local controls in stage 1, the desired precision being set to ε = 0.10 (n=19 maximum).

Number of subjects required 60 patients with significant uptake on FDG-PET imaging after neo-adjuvant chemotherapy (75 pre-inclusion) will be included. Only half of these 60 patients (30) are expected to be definitely eligible with F-miso PET identifying hypoxic areas. Out these 30 eligible patients, we assume that 5 will not be evaluable, so that a total of 25 evaluable patients will be assessable.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage III non-small-cell lung cancer candidate for curative radio-chemotherapy
* The final inclusion is granted after completion of a dosimetric study confirming that the dose objectives (minimum dose of 60 Gy in 99% of target volume) and constraints to organs at risk can be achieved.

Exclusion Criteria:

* Other cancer
* no evaluable tumor target
* Absence of binding to FDG-PET tests before primary chemotherapy
* Patients for which radiotherapy with curative intent is not indicated
* History of neoplastic disease of less than 5 years or progressive
* Patient already included in another clinical trial
* Pregnant, likely to be or during breastfeeding
* performance index OMS ≥2
* Indicating renal insufficiency against Cisplatin treatment
* Protected adults
* Unable to submit to medical study for reasons geographical, social or physical
* Patients with poorly controlled diabetes blood sugar ≥10 mmol/L
* hypersensitivity to FDG or any excipients of the radiopharmaceutical
* hypersensitivity to Fmiso or any excipients of the radiopharmaceutical
* Patients unable to understand the study (language ...)
* Patients not affiliated to the "sécurité social"

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-03 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of local control | 3 month
  to evaluate the rate of local control after dose complement in hypoxic lesions [maximum dose without the fraction of total lung volume receiving more that 20 Gy exceeding 30% of the lung (V20)], as determined by F-miso PET/CT.

SECONDARY OUTCOMES:
3 months and 1 year toxicity | 1 year
  3 months and 1 year toxicity measured according CTCAE 4.0
Percentage of patients for whom the RT dose could be increased | 3 years
  Percentage of patients for whom the RT dose could be increased
Simultaneous variation of the glucose metabolism and hypoxia during radiotherapy | 3 years
  comparaison of both exam PETscan FDG and PETscan FMISO performed during radiotherapy
Predictive value on 1-year survival | 1 year
  Predictive value on 1-year survival probability of the variations in glucose metabolism and hypoxia during radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Henri Becquerel, Rouen, France

REFERENCES:
- [Derived] Ganem J, Thureau S, Gardin I, Modzelewski R, Hapdey S, Vera P. Delineation of lung cancer with FDG PET/CT during radiation therapy. Radiat Oncol. 2018 Nov 12;13(1):219. doi: 10.1186/s13014-018-1163-2. PMID 30419929
- [Derived] Thureau S, Dubray B, Modzelewski R, Bohn P, Hapdey S, Vincent S, Anger E, Gensanne D, Pirault N, Pierrick G, Vera P. FDG and FMISO PET-guided dose escalation with intensity-modulated radiotherapy in lung cancer. Radiat Oncol. 2018 Oct 23;13(1):208. doi: 10.1186/s13014-018-1147-2. PMID 30352608
- [Derived] Vera P, Thureau S, Chaumet-Riffaud P, Modzelewski R, Bohn P, Vermandel M, Hapdey S, Pallardy A, Mahe MA, Lacombe M, Boisselier P, Guillemard S, Olivier P, Beckendorf V, Salem N, Charrier N, Chajon E, Devillers A, Aide N, Danhier S, Denis F, Muratet JP, Martin E, Riedinger AB, Kolesnikov-Gauthier H, Dansin E, Massabeau C, Courbon F, Farcy Jacquet MP, Kotzki PO, Houzard C, Mornex F, Vervueren L, Paumier A, Fernandez P, Salaun M, Dubray B. Phase II Study of a Radiotherapy Total Dose Increase in Hypoxic Lesions Identified by 18F-Misonidazole PET/CT in Patients with Non-Small Cell Lung Carcinoma (RTEP5 Study). J Nucl Med. 2017 Jul;58(7):1045-1053. doi: 10.2967/jnumed.116.188367. Epub 2017 Mar 2. PMID 28254869